CLINICAL TRIAL: NCT06759103
Title: Electronic Archive of Patients With Diagnosis and Suspected Prenatal Diagnosis of Aortic Coarctation
Acronym: ACOAP
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ACOAP
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Aortic Coarctation
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prosective and retrospective observational study is to analyze the clinical and echocardiographic characteristics of infants with prenatal diagnosis of suspected aortic coarctation (CoAo) in order to identify clinical and instrumental elements that can predict the risk of developing aortic coarctation in the neonatal period so that we can identify patients who are at high risk and would therefore require intensive care and observation; compared with low-risk patients, for whom early discharge would be evaluable.

DETAILED DESCRIPTION:
Our study has the intention of analysing the clinical and echocardiographic characteristics of infants with prenatal and neonatal diagnosis of suspected CoAo, transferred at birth to the O.U. of Cardiology and Paediatric Cardiac Surgery at the Policlinico di Sant' Orsola in order to identify reliable predictors of CoAo, in particular reliable in presence of the ductus arteriosus of Botallo.

It is an observational study: patients participating in the study will not undergo to any procedures outside the normal clinical practice; likewise, the clinical variables that will be collected for study are those that are commonly collected by the physician in daily clinical practice. This study therefore involves the observation of current clinical practice without the application of any kind of 'intervention'.The primary objective of the study is:

to identify the clinical and/or echocardiographic features predictive of the development of Aortic Coarctation through the creation of a data collection with which to census all patients with a diagnosis of suspected or overt Aortic Coarctation, admitted from 01/01/2007 to 31/12/2026 at the Paediatric Cardiology and Cardiac Surgery Centre of the Policlinico di Sant'Orsola, Bologna.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre-natal or post-natal diagnosis of aortic coarctation from 01 January 2000 until approval (retrospective phase) and from approval until 31 December 2026 (prospective phase)

Exclusion Criteria:

* Patients whose diagnosis of aortic coarctation is postnatal, considered to be >1 month after birth
* prenatal diagnosis of genetic disease (e.g., Turner's Sdr)
* coarctation in the setting of complex congenital heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected prenatal diagnosis of aortic coarctation, referred to our next center from 01 January 2000 to 31 December 2026 will be considered going to include, according to a preliminary analysis, a cohort of about 150 patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify clinical or echocardiographic features, predictive of development of aortic coarctation | Through study completion, an average of 5 years
  The study is observational, non-interventional in nature. Patients will be treated according to clinical practice. In particular, information will be collected regarding:
  * ECG
  * Transthoracic echocardiogram
  * Interventional or surgical procedures
  * Follow-up examinations
  The diagnosis of isthmic aortic coarctation is based on the echocardiographic finding. Clinically, coarctation is defined as significant and with indication for surgical correction in the presence of signs of reduced abdominal systemic perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ylenia Bartolacelli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No